CLINICAL TRIAL: NCT02943187
Title: Novel Functional Medicine Intervention With Cognitive Training for Mild Cognitive Impairment (MCI): A Multiple Baseline Study Across Cases
Brief Title: Multidisciplinary Intervention for Mild Cognitive Impairment
Acronym: (MCI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gibson Institute of Cognitive Research (Industry)
Collaborators: True Life Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GICR-1012
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutrition and Cognitive Training (Experimental): The intervention includes a physician-directed diet, exercise, and nutritional supplementation regimen, combined with a 60-hour, clinician-delivered cognitive training program created by LearningRx.
  Interventions: Behavioral: Cognitive training; Dietary Supplement: Nutrition

INTERVENTIONS:
Behavioral: Cognitive training — A clinician will deliver three 90-minute cognitive training sessions per week for 14 weeks. There are 16 different categories of leveled training procedures sequenced in intensity and difficulty for a total of 530 training tasks.
Dietary Supplement: Nutrition — Participants will be given dietary recommendations and nutritional supplements to optimize cognition.

SUMMARY:
The purpose of this investigation is to conduct a series of case studies on the impact of a novel functional medicine approach to improving cognitive skills, brain structure, and daily functioning for participants with Mild Cognitive Impairment (MCI).

DETAILED DESCRIPTION:
Using a multiple baseline design across cases with start point randomization, the proposed study will examine the outcomes from a combination of optimized diet, exercise, nutritional supplements, and cognitive training across domains on standardized measures used to monitor treatment effectiveness for Mild Cognitive Impairment (MCI).

ELIGIBILITY:
Inclusion Criteria:

* Age 50+ previously diagnosed with MCI
* Living in the greater Colorado Springs area

Exclusion Criteria:

* No braces, metal implants, or claustrophobia that would contraindicate magnetic resonance imaging

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-10; Primary Completion 2018-12 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Evidence of overall cognitive function improvement | within 14 days after completing the intervention
  Confirmed by change in pretest to post-test scores on the Dementia Rating Scale (DRS-2)

SECONDARY OUTCOMES:
Evidence of improvement in executive function | within 14 days after completing the intervention
  As confirmed by pretest to post-test changes on the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A)
Evidence of improvement in cognitive flexibility | within 14 days after completing the intervention
  As confirmed by pretest to post-test changes on a Trail Making Test
Evidence of change in brain function | within 30 days after completing the intervention
  Confirmed by change in pretest to post-test neuroimaging using MRI
Evidence of improvement in visual attention | with 14 days after completing the intervention
  Confirmed by change in pretest to post-test scores on the Conners Continous Performance Test (CPT-3)
Evidence of improvement in auditory attention | with 14 days after completing the intervention
  Confirmed by change in pretest to post-test scores on the Auditory Attention Test (CATA)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Ledbetter, PhD, Principal Investigator — Gibson Institute of Cognitive Research; Amy L Moore, PhD, Study Director — Gibson Institute of Cognitive Research; Randolph James, MD, Principal Investigator — True Life Medicine; Dick M Carpenter, PhD, Principal Investigator — University of Colorado, Colorado Springs
Locations (1):
- Gibson Institute of Cognitive Research, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Harvard Dataverse

REFERENCES:
- [Result] James, R., Moore, A.L., Carpenter, D., Miller, T., & Ledbetter, C. (2019). Feasibility of a Functional Medicine Approach to Slowing Clinical Cognitive Decline in Patients Over Age 55: A Multiple Case Study Report. OBM Integrative and Complementary Medicine, 4(3). doi: 10.21926/obm.icm.1903054 Retrieved from https://www.lidsen.com/journals/icm/icm-04-03-054
- See also: James et al study link — https://www.lidsen.com/journals/icm/icm-04-03-054